CLINICAL TRIAL: NCT03422848
Title: Hydration to Optimize Metabolism
Acronym: H2O-metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Olle Melander, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016894
Record Dates: First submitted 2018-01-06; First posted 2018-02-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Glucose, High Blood
Keywords: hydration; water; vasopressin; copeptin; glucose; OGTT; insulin; glucagon
MeSH Terms: conditions — Diabetes Insipidus; Insulin Resistance | interventions — Water

STUDY DESIGN:
Intervention Model Description: Parallel-group RCT with two arms during 12 months. Subjects will be randomized to the water-intervention (in total 1.5 L increment daily on the top of habitual intake) and control groups (1:1) by computer-generated block randomization. Both groups will receive general life style advice (general oral and written advice on diet and physical activity).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water intervention arm (Active Comparator): The water intervention group will increase their habitual daily water intake with 1.5 L of tap water. Furthermore they will receive general life style advice (general oral and written advice on diet and physical activity).
  Interventions: Dietary Supplement: Water; Behavioral: general life style advice
- Control arm (Other): Control group that will receive general life style advice (general oral and written advice on diet and physical activity).
  Interventions: Behavioral: general life style advice

INTERVENTIONS:
Dietary Supplement: Water — Increased daily water intake with 1.5 L of water on top of habitual water intake.
  Arms: Water intervention arm
Behavioral: general life style advice — oral and written advice on diet and physical activity

SUMMARY:
This study evaluates hydration (1.5 L of water daily during 1 year) in the lowering of blood glucose concentration in adults with signs of dehydration (elevated levels of the vasopressin marker copeptin and high urine osmolality). Half of participants will in addition to lifestyle advice receive extra water on top of their habitual fluid intake, and the other half (control) will receive only lifestyle advice.

DETAILED DESCRIPTION:
High plasma concentration of vasopressin (i.e. antidiuretic hormone) is a novel and independent risk factor for type 2 diabetes, the metabolic syndrome, cardiovascular disease and premature death. The main physiological role of vasopressin is to maintain constant plasma osmolality. Previous studies in rats and mendelian randomization studies in humans suggest causality between elevated vasopressin concentration and elevated plasma glucose concentration. As vasopressin can be suppressed by increasing water intake, we hypothesize that water supplementation in individuals with high vasopressin can lower plasma glucose and prevent diabetes.

The aim of this project is to test in a single-centre randomized clinical trial (RCT), if water supplementation in subjects with high plasma levels of vasopressin (measured by a stable vasopressin marker of its precursor hormone called copeptin) can reduce fasting levels of glucose (primary outcome measure), risk of new-onset diabetes and other cardiometabolic risk factors (secondary outcome measures).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent, age 20-75 years with high plasma concentration of vasopressin (plasma concentration of copeptin of > 6.1 pmol/L in women and > 10.7 pmol/L in men) and 24 hour urine osmolality > 600 milliosmol (mOsm) /kg water.

Exclusion Criteria:

* 24 hour urine volume > 1.5 L, pregnancy or breastfeeding, plasma sodium < 135 mmol/L, use of diuretics, lithium or selective serotonin reuptake inhibitor (SSRI) drugs, chronic kidney disease (estimated glomerular filtration rate < 30 mL/min), heart failure, inflammatory bowel disease, type 1 diabetes or type 2 diabetes treated with insulin, vulnerable subjects (subjects with legal guardian, with loss of personal liberty).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose concentration (mmol/L) | 12 months
  Difference in change of fasting plasma glucose between water intervention arm and control arm.

SECONDARY OUTCOMES:
Diabetes incidence | 12 months
  Difference in diabetes incidence between water intervention arm and control arm.
Post oral glucose load glucose concentration (mmol/L) | 12 months
  Difference in change of post oral glucose load glucose concentration (mmol/L) between water intervention arm and control arm
Fasting insulin concentration (mIE/L) | 12 months
  Difference in change of fasting insulin (mIE/L) between water intervention arm and control arm
Post oral glucose load insulin concentration (mIE/L) | 12 months
  Difference in change of post oral glucose load insulin concentration (mIE/L) between water intervention arm and control arm
Fasting glucagon concentration (pmol/L) | 12 months
  Difference in change of fasting glucagon (pmol/L) between water intervention arm and control arm
Post oral glucose load glucagon concentration (pmol/L) | 12 months
  Difference in change of post oral glucose load glucagon concentration (pmol/L) between water intervention arm and control arm
HbA1c concentration (mmol/mol) | 12 months
  Difference in change of HbA1c (mmol/mol) between water intervention arm and control arm
Waist circumference (cm) | 12 months
  Difference in change of waist circumference (cm) between water intervention arm and control arm
Body mass index (kg/m^2) | 12 months
  Difference in change of body mass index (kg/m^2) between water intervention arm and control arm
Systolic blood pressure (mmHg) | 12 months
  Difference in change of systolic blood pressure (mmHg) between water intervention arm and control arm
Diastolic blood pressure (mmHg) | 12 months
  Difference in change of diastolic blood pressure (mmHg) between water intervention arm and control arm
Triglyceride concentration (mmol/L) | 12 months
  Difference in change of triglycerides (mmol/L) between water intervention arm and control arm
HDL cholesterol concentration (mmol/L) | 12 months
  Difference in change of HDL cholesterol (mmol/L) between water intervention arm and control arm
LDL cholesterol concentration (mmol/L) | 12 months
  Difference in change of LDL cholesterol (mmol/L) between water intervention arm and control arm
Apolipoprotein B concentration (g/L) | 12 months
  Difference in change of Apolipoprotein B (g/L) between water intervention arm and control arm
Apolipoprotein A1 concentration (g/L) | 12 months
  Difference in change of Apolipoprotein A1 (g/L) between water intervention arm and control arm
Urine albumin/creatinine ratio (g/mol) | 12 months
  Difference in change of urine albumin/creatinine ratio (g/mol) between water intervention arm and control arm
Estimated glomerular filtration rate (mL/min/1,73 m2) | 12 months
  Difference in change of estimated glomerular filtration rate (mL/min/1,73 m2) between water intervention arm and control arm
Creatinine clearance (mL/min) | 12 months
  Difference in change of creatinine clearance (mL/min) between water intervention arm and control arm
Fasting cortisol concentration (nmol/L) | 12 months
  Difference in change of fasting cortisol (nmol/L) between water intervention arm and control arm
Fasting adrenocorticotropic hormone concentration (pmol/L) | 12 months
  Difference in change of fasting adrenocorticotropic hormone (pmol/L) between water intervention arm and control arm
C-reactive protein concentration (mg/L) | 12 months
  Difference in change of C-reactive protein (mg/L) between water intervention arm and control arm
Hair cortisol concentration (pg/mg) | 12 months between samplings
  Difference in change of hair cortisol (pg/mg) between water intervention arm and control arm. Hair cortisol is a measure of chronic stress exposure 3 months prior to sampling.

OTHER OUTCOMES:
Fasting plasma glucose concentration in pre-specified subgroups | 12 months
  glucose reduction in A) subjects who remain high in copeptin from population screening to main study baseline, B) subjects with the highest (top tertile) baseline copeptin, C) subjects with/without diabetes mellitus at baseline, D) subjects with/without impaired fasting glucose (diabetes+impaired/not impaired), E) men and women separately.

CONTACTS AND LOCATIONS:
Overall Officials: Olle Melander, M.D., Prof., Principal Investigator — Lund University
Locations (1):
- KFE, Skåne University Hospital in Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03422848/Prot_000.pdf
  • Statistical Analysis Plan: Original Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03422848/SAP_001.pdf
  • Statistical Analysis Plan: Detailed Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03422848/SAP_002.pdf